CLINICAL TRIAL: NCT05025904
Title: The Functional Mechanism of the Neurovascular Coupling: an fMRI-EEG Study in Depressive Depression
Brief Title: Real-time fMRI Neurofeedback for Mild/Moderate Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Research Center of Fundamental and Translational Medicine, Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-15-00183
Record Dates: First submitted 2021-08-18; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Depression Mild; Depression Moderate
Keywords: Neurofeedback; Functional Magnetic Resonance Imaging; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of 3 groups: real-time fMRI neurofeedback (rt-fMRI NFB), EEG neurofeedback (aborted), and cognitive behavioral therapy (CBT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real-time fMRI neurofeedback (rt-fMRI NFB) (Experimental): The duration of a session was approximately a half-hour. The course duration was 8 sessions. The preferred frequency was once a week, however, the schedule was flexibly adjusted for patients' convenience.
  Interventions: Behavioral: Real-time fMRI neurofeedback (rt-fMRI NFB)
- Сognitive behavioral therapy (CBT) (Active Comparator): The duration of a session was approximately an hour/hour and a half. The course duration was 8 individual and 8 group sessions and included home assignments. The preferred frequency was twice a week, however, the schedule was flexibly adjusted for patients' convenience and for improving benefits of the treatment.
  Interventions: Behavioral: Сognitive behavioral therapy (CBT)
- EEG neurofeedback (EEG NFB) (Active Comparator): The duration of a session was approximately a half-hour. The course duration was 16 sessions. The preferred frequency was twice a week, however, the schedule was flexibly adjusted for patients' convenience.
  Group was preliminarily aborted for lack of time and participants in order to assign more patients to the abovementioned arms.
  Interventions: Behavioral: EEG neurofeedback (EEG NFB)

INTERVENTIONS:
Behavioral: Real-time fMRI neurofeedback (rt-fMRI NFB) — Real-time fMRI neurofeedback targeting control of the left medial prefrontal cortex. Participants continuously received visual feedback on the level of activity within the 2D region of interest corrected to the whole-slice brain volume activity. Up- and downregulation blocks were switched for better control.
  Arms: Real-time fMRI neurofeedback (rt-fMRI NFB)
Behavioral: Сognitive behavioral therapy (CBT) — A combination of individual and small-group cognitive behavioral therapy by an experienced medical psychologist and a psychiatrist.
  Arms: Сognitive behavioral therapy (CBT)
Behavioral: EEG neurofeedback (EEG NFB) — EEG neurofeedback targeting frontal alpha asymmetry index. Participants continuously received visual feedback on their frontal alpha asymmetry index. Up-regulation condition only was utilized.
  Arms: EEG neurofeedback (EEG NFB)

SUMMARY:
The aim of the study is to compare the effects of the self-regulation (neurofeedback) of the fMRI signal of the prefrontal cortex in depression to ones of more conventional non-pharmacological treatment, primarily, psychotherapy.

DETAILED DESCRIPTION:
The study was devoted to the neural, clinical, and psychological effects of the rt-fMRI neurofeedback for mild/moderate depression. Recruited unmedicated patients suffering from depression were assigned either to the fMRI neurofeedback (8 sessions of the left prefrontal cortex activity regulation) or to the active control group, i.e., a double dosage of cognitive-behavioral treatment or EEG neurofeedback (preliminary aborted). Depression symptoms were measured at baseline, at mid-treatment, and at post-treatment points. Some inventories of depression and related traits were also given. In the rt-fMRI group, self-regulation learning was also estimated by means of the fMRI signal change.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of unipolar depressive disorder on ICD-10 (F32, F33, F34.1)
* Sufficient self-regulation ability (verified with 3 sessions of ALAY EEG neurofeedback)

Exclusion Criteria:

* Serious somatic, mental, or substance abuse problem other than depression
* Depression secondary to other mental or somatic conditions
* Psychotic features in depression or comorbid psychotic disorder
* Serious suicide risk
* Seasonal depression
* Receiving or planning to receive psychotropic medications
* Receiving cardiovascular medications
* General MRI exclusions
* Current pregnancy
* IQ<70 (established with Raven's progressive matrices)
* Previous experience with neurofeedback

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Change in depression symptoms severity from baseline to end-treatment | 4.5 months on average
  Montgomery-Asberg Depression Rating Scale (MADRS), scores ranging 0-54, higher scores indicate more severe depression
Change in depression symptoms severity from baseline to mid-treatment | 2.5 months on average
  Montgomery-Asberg Depression Rating Scale (MADRS), scores ranging 0-54, higher scores indicate more severe depression

SECONDARY OUTCOMES:
Change in subjective depression severity, test 1 from baseline to end-treatment | 4.5 months on average
  Beck Depression Inventory (BDI), scores ranging 0-63, higher scores indicate more severe subjective depression
Change in subjective depression severity, test 1 from baseline to mid-treatment | 2.5 months on average
  Beck Depression Inventory (BDI), scores ranging 0-63, higher scores indicate more severe subjective depression
Change in subjective depression severity, test 2 from baseline to end-treatment | 4.5 months on average
  Zung Self-Rating Depression Scale (ZSRDS), scores ranging 20-80, higher scores indicate more severe subjective depression
Change in subjective depression severity, test 2 from baseline to mid-treatment | 2.5 months on average
  Zung Self-Rating Depression Scale (ZSRDS), scores ranging 20-80, higher scores indicate more severe subjective depression
Change in the raw estimate of subjective depression severity from baseline to end-treatment | 4.5 months on average
  Hospital Anxiety and Depression Scale (HADS), depression subscale, scores ranging 0-21, higher scores indicate more severe subjective depression
Change in the raw estimate of subjective depression severity from baseline to mid-treatment | 2.5 months on average
  Hospital Anxiety and Depression Scale (HADS), depression subscale, scores ranging 0-21, higher scores indicate more severe subjective depression

OTHER OUTCOMES:
Change in adult anxious attachment from baseline to end-treatment | 4.5 months on average
  Experience in Close Relationships (ECR), anxious attachment subscale, scores ranging 15-105, higher scores indicate more attachment disruption
Change in adult anxious attachment from baseline to mid-treatment | 2.5 months on average
  Experience in Close Relationships (ECR), anxious attachment subscale, scores ranging 15-105, higher scores indicate more attachment disruption
Change in adult avoidant attachment from baseline to end-treatment | 4.5 months on average
  Experience in Close Relationships (ECR), avoidant attachment subscale, scores ranging 15-105, higher scores indicate more attachment disruption
Change in adult avoidant attachment from baseline to mid-treatment | 2.5 months on average
  Experience in Close Relationships (ECR), avoidant attachment subscale, scores ranging 15-105, higher scores indicate more attachment disruption
Change in rumination level from baseline to end-treatment | 4.5 months on average
  Rumination Response Scale (RRS), total rumination score, scores ranging 22-88, higher scores indicate more rumination
Change in rumination level from baseline to mid-treatment | 2.5 months on average
  Rumination Response Scale (RRS), total rumination score, scores ranging 22-88, higher scores indicate more rumination
Change in alexithymia level from baseline to end-treatment | 4.5 months on average
  Toronto Alexithymia Scale (TAS-26), scores ranging 26-130, higher scores indicate more alexithymia
Change in alexithymia level from baseline to mid-treatment | 2.5 months on average
  Toronto Alexithymia Scale (TAS-26), scores ranging 26-130, higher scores indicate more alexithymia

CONTACTS AND LOCATIONS:
Overall Officials: Mark B. Shtark, Ph.D., Study Director — FRC FTM
Locations (1):
- Federal Reserch Center of Fundamental and Translational Medicine, Novosibirsk, Russia